CLINICAL TRIAL: NCT03195309
Title: A Comparison of Different Concentration Ropivacaine Combination With Fentanyl for Patient-controlled Epidural Analgesia After Cesarean Delivery
Brief Title: A Comparison of Different Concentration Ropivacaine for Patient-controlled Epidural Analgesia
Acronym: PCEA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(1)-20160019
Record Dates: First submitted 2017-04-18; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-04

CONDITIONS: Epidural Anesthesia; Cesarean Section
Keywords: Cesarean Delivery; Ropivacaine; Fentanyl; Patient-controlled Epidural Analgesia
MeSH Terms: interventions — Ropivacaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: All patients were received epidural anesthesia with 2% Lidocaine and patient-controlled epidural analgesia (PCEA) for post- operative pain control. PCEA randomly allocated into three groups. Group A patients received 0.08% ropivacaine plus 4 mcg /mL fentanyl, Group B patients received 0.08% ropivacaine plus 2mcg /mL fentanyl, and Group C patients received 0.16 % ropivacaine plus 2 mcg /mL fentanyl. Dermographic data, dosage of PCEA during first 48 hours post-operation，NRS scores, patient satisfaction and the intensity of motor block will be recorded and analyzed.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant do not know which formula they are receive. Nor do the daily care providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Active Comparator): Group A patients received 0.08% ropivacaine plus 4 mcg /mL fentanyl
  Interventions: Drug: Ropivacaine; Drug: Fentanyl
- Group B (Active Comparator): Group B patients received 0.08% ropivacaine plus 2mcg /mL fentanyl
  Interventions: Drug: Ropivacaine; Drug: Fentanyl
- Group C (Active Comparator): Group C patients received 0.16 % ropivacaine plus 2 mcg /mL fentanyl
  Interventions: Drug: Ropivacaine; Drug: Fentanyl

INTERVENTIONS:
Drug: Ropivacaine — Compare different concentration of ropivacaine and fentanyl for elective Cesarean delivery post operative pain control.
  Other Names: Ropica
Drug: Fentanyl — Compare different concentration of ropivacaine and fentanyl for elective Cesarean delivery post operative pain control.

SUMMARY:
To compare the postoperative analgesic effect and the intensity of motor block in different concentration ropivacaine plus fentanyl when used epidurally with a patient-controlled analgesia device after Cesarean delivery.

DETAILED DESCRIPTION:
1. Written informed consent must be obtained before any study specific procedures are undertaken.
2. All patients were received epidural anesthesia with 2% Lidocaine and patient-controlled epidural analgesia (PCEA) for post- operative pain control. PCEA randomly allocated into three groups. Group A patients received 0.08% ropivacaine plus 4 mcg /mL fentanyl, Group B patients received 0.08% ropivacaine plus 2mcg /mL fentanyl, and Group C patients received 0.16 % ropivacaine plus 2 mcg /mL fentanyl. Dermographic data, dosage of PCEA during first 48 hours post-operation，NRS scores, patient satisfaction and the intensity of motor block will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Female undergoing elective Cesarean delivery and receive patient-controlled epidural analgesia

Exclusion Criteria:

* With the comorbidity of chronic heart, lung, liver and renal disease, chronic alcoholism, allergy to ropivacaine, poor epidural function and combine other anesthesia method

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only include pregnant female receiving elective Cesarean delivery and post-operative epidural analgesia
Enrollment: 120 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores on the numeric rating scale | The investigators measured numeric score changing at 5 different timing. The first is when arrival post-operative care unit, the second is when arrival post-operative care unit for 2 hours. And then 6,24,48 hours after operation.
  The investigators use numeric rating scale(0~10) for pain severity measurement, 0 for no pain, 10 is the most severe pain

SECONDARY OUTCOMES:
Change From Baseline in Patient satisfaction scale | The investigators measured numeric score changing at 5 different timing. The first is when arrival post-operative care unit, the second is when arrival post-operative care unit for 2 hours. And then 6,24,48 hours after operation.
  Patient satisfaction scale (1~4), 1 for very satisfied, 2 for satisfied, 3 for fair, and 4 for unsatisfied

OTHER OUTCOMES:
Change From Baseline in modified Bromage scale | The investigatorsmeasured numeric score changing at 5 different timing. The first is when arrival post-operative care unit, the second is when arrival post-operative care unit for 2 hours. And then 6,24,48 hours after operation.
  The investigators use modified Bromage scale for motor block evaluation. Modified Bromage scale(0~3), 0 for no motor block. 1 for inability to raise extended leg, able to move knees and feet. 2 for inability to raise extended leg and move knee, able to move feet. 3 for complete block of motor limb

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Fang Huang, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No